CLINICAL TRIAL: NCT03923712
Title: Effect of Supervised Physical Exercise on Brain, Cognition, OMICs, Molecular Markers and Functional Status in Older People at Risk of Mild Cognitive Impairment: Rationale, Design and Methodology.
Brief Title: Exercise, Brain, Cognition, OMICs, Molecular Markers and Functionality in People at Risk of Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Collaborators: Centro de Excelencia en Metabolómica y Bioanálisis (CEMBIO) (Unknown); Servicio Central de Neuroimagen de la Universidad Pablo de Olavide (Unknown); Consejería de Salud y Bienestar Social, Andalucía (Unknown)
Responsible Party: Principal Investigator, David Jimenez Pavon, Ramón y Cajal Senior Researcher, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DEP2016-76123-R; PI-0002-2017 (Other Grant/Funding Number: Fondos FEDER-ITI, Junta de Andalucia)
Record Dates: First submitted 2018-06-01; First posted 2019-04-23 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Mild Cognitive Impairment; Alzheimer Dementia
Keywords: Physical exercise; ageing; dementia; Alzheimer; magnetic resonance image; cerebral; cognition; metabolomic; older people; mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Motor Activity; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants randomly assigned to control group will be instructed to maintain their normal life habits with respect to physical activity and diet. During the 5 months of intervention participants from this group will receive at least one call from the researchers to be interested in their health status and inform them about the next evaluation appointment, as well as, an objectively evaluation of the main behaviours in the middle of intervention. Investigators will inform about the relevance of attending the full process and respecting the condition and rule as control. Participants from the control group will be freely offered the possibility to get involve in a similar intervention protocol at the end of the study in order to benefit from the potential positive effect of exercise.
- Supervised exercise programme (Experimental): 5 months of supervised physical exercise program. The individualized and progressive Health periodization model will be applied establishing an initial individualizing period, as well as identifying any need or adaptation to apply during the exercise program. The physical exercise program will be applied in a period of progressive increase whose initial objective will be to reach the volume and intensity established by the international recommendations of physical activity (http://www.health.gov/paguidelines/) for this population. Briefly, a volume of 150 min/week of moderate-vigorous physical activity (60% -85% reserve heart rate) spread over a maximum of 5 days and including force work 2-3 days/week. The training load will progressively increase with a wave and flexible periodization.
  Interventions: Behavioral: Supervised Exercise Programme

INTERVENTIONS:
Behavioral: Supervised Exercise Programme — The methodology will be multicomponent, including aerobic, strength, coordination-cognitive and balance-agility. The physical exercise sessions will be designed in such a way that they work the dimensions but being attractive and motivating for the participants. Each session will include 10 minutes of warm-up with smooth running and mobility exercises; 35-40 minutes of aerobic, strength, coordination-cognitive and balance-agility progressively developed; and 10 minutes back to calm at low intensity with stretching exercises. Nutritional intervention will not be included. For quality purposes, we will use small groups (10-15 pers). After each session participants will be asked about their subjective perception of the effort and the intensity will be controlled by heart rate monitors.
  Arms: Supervised exercise programme

SUMMARY:
This project aims to examine the effect of a 5-month period supervised exercise intervention on brain, cognition, OMICs, Molecular Markers and functional status in older people at risk of mild cognitive impairment. Secondarily, the effect of this intervention on antioxidant capacity, lipid metabolism and glucose, physical health (functional capacity, blood pressure, body composition) and mental (quality of life and depression) will be studied, as well as other factors risk (genetic and biological) for the development of Alzheimer. A total of 100 people aged between 65 and 75 years old at risk of mild cognitive impairment will be randomly distributed in the supervised exercise intervention group (n = 50) and control group (n = 50). The design will include a 5-month intervention with measurements at pre and post intervention and a third measurement (retest) after 3 months of completion. The multicomponent supervised exercise program will include aerobic, strength, cognitive and coordinative-agility-balance works, and progression will be established in different load parameters (frequency, volume, intensity, density). Therefore, randomized controlled studies are needed to know the specific effect of dose-response considering the various dimensions in parallel such as neuroimaging, cognitive status and OMICS. This will allow us to understand from a comprehensive perspective the causes and mechanisms underlying the response. This project will significantly increase scientific knowledge about the role of exercise on brain as a therapeutic measure in people at risk of mild cognitive impairment from a multidimensional perspective. The project will have a significant impact at social and economic level by transferring the study findings to social and health setting by means of agents and networks provided for the project.

ELIGIBILITY:
Inclusion Criteria:

* Do not present any physical illness that prevents you from doing physical activity
* Able to communicate without problems
* Able to read and understand informed consent as well as the object of the study

Exclusion Criteria:

* Acute or terminal illness
* Diagnosis of Alzheimer's
* History of cranioencephalic trauma with loss of consciousness
* History of cerebral infarction, epilepsy, brain tumor
* Unstable cardiovascular disease
* Recent fracture in upper or lower limb
* Alcohol abuse and / or habitual drug use or drug infusion pump
* Presence of pacemakers, defibrillator, metallic implants in the head, intraocular and / or maxillo-facial structures, dental prostheses incompatible with magnetic resonance studies
* Intravascular devices (stent, Coil, filter), heart valve, aneurysm clip, neurostimulator, intravascular catheter with metal or cardiovascular bypass
* Severe visual or auditory problems, implant in the middle / inner ear
* Do not want to complete the study or be assigned to the control group
* He/she is participating in another research study that may influence the present project.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Assessed changes from Baseline Neuroimaging Markers of Brain Structures (thickness in mm; volumes in mm) | up to 24 weeks
  Brain magnetic resonance images will be acquired in a Philips-Ingenia 3-Tesla scanner with a 32-channel digital coil exclusively dedicated to skull (Philips, The Netherlands) with the anatomical sequences:
  1. Sequence T1-3D in sagittal orientation. This sequence will quantify the cortical thickness and perform morphometric studies of cortical and subcortical structures.
  The pattern of cortical thickness changes and the volume of different brain structures will be obtained with the tools implemented in the software Freesurfer v5.3 and SPM12.
Assessed changes from Baseline Neuroimaging Markers of Brain Function (level of activity in percentage) | up to 24 weeks
  Brain magnetic resonance images will be acquired in a Philips-Ingenia 3-Tesla scanner with a 32-channel digital coil exclusively dedicated to skull (Philips, The Netherlands) with the anatomical sequences:
  1. DTI (Diffusion Tensor Imaging) sequence in axial orientation. This sequence will allow to evaluate the properties of the microstructure of the white matter and its nerve fiber tracts.
  2. T2 / FLAIR sequences in axial orientation. Both sequences will be used to determine the degree of involvement of the deep and periventricular white matter using the Fazekas scale.
Assessed changes from Baseline Cognitive Status | up to 36 weeks
  An overall SCORE (z-score values or similar;higher value for better outcome) of the 8 measurements on cognitive status will be developed to arrive at one reported value:
  1. - Clinical Dementia Rating -CDR: This is a valid and reliable instrument for staging dementia.
  2. - Mini Mental State Examination to detect cognitive deterioration.
  3. - Trail Making Test -TMT: This is an indicator of the speed of cognitive processing and executive functioning. 2 parts.
  4. - Boston Naming Test to assess the ability to name objects.
  5. - Clock Drawing Test -CDT: valid test for evaluation of cognitive deterioration.
  6. - Rey Auditory Verbal Learning Test -RAVLT: learning and verbal episodic memory.
  7. - The Stroop Color and Word Test -SCWT: examines basic psychological processes (cognitive flexibility, selective attention, resistance to interference from external stimuli and cognitive inhibition).
  8. -Controlled Oral Word Association Test -COWAT: designed to assess verbal fluency.
Assessed changes from Baseline OMICs Analysis | up to 36 weeks
  To carry out the analysis of the OMICs a full untargeted profiling will be carried out in the pre and post-intervention and retest measurements for different OMICS including metabolomics, proteomics,etc. For these analyzes, the following large equipment and techniques will be used, ultrahigh performance liquid chromatography / mass spectrometry (LC-quadrupole-time of flight, QTPF-MS, Agilent 1200-Agilent 6520); capillary electrophoresis / mass spectrometry (CE, TOF-MS, Agilent 7100-Agilent 6210) and gas chromatography / mass spectrometry (GC, EI-GC), mass spectrometry (capillary electrophoresis / mass spectrometry, CE-TOF-MS; Q-MS, (Quadrupolo, Agilent 7890A-Agilent 5965C) In addition, data processing platforms will be used, both mass databases and statistical tools for multivariate analysis: Mass Hunter, Mass Profiler Professional, SIMCA, MATLAB.
Assessed changes from Baseline Molecular Makers | up to 36 weeks
  The telomere length will be measured by quantitative real-time PCR (RT-qPCR) following the method previusly described. Briefly, the DNA from the cell fraction of the blood will be extracted with the DNeasy Blood & Tissue Kit (Qiagen) following the manufacturer's specifications. The DNA concentration of the sample, as well as its integrity, will be confirmed in a NanoDrop 2000. For the RT-qPCR the telomeric sequence will be amplified as well as a single copy gene sequence to normalize. Calibration curves will be made with serial dilutions of known concentration of both the gene sequence as well as an oligo specially designed to contain 114 copies of the TTAGGG telomeric sequence. The RT-qPCR will be carried out with 20 ng of DNA using myScript SYBR Green PCR Kit (ROCHE). The PCR conditions are: 10 min at 95 ° C, followed by 40 cycles of 95 ° C for 15 sec and 60 ° C for 1 min, followed by the corresponding dissociation curve.

SECONDARY OUTCOMES:
Assessed changes from Baseline Physical Health Parameters on Functional capacity: Muscle-skeletal | up to 36 weeks
  Consist in a Standardized field test battery including:
  1.Muscle-skeletal (number of repetitions)
Assessed changes from Baseline Physical Health Parameters on Functional capacity: Cardiorespiratory fitness | up to 36 weeks
  Consist in a Standardized field test battery including:
  2.Cardiorespiratory fitness (metres and estimated maximal oxygen uptake-VO2max)
Assessed changes from Baseline Physical Health Parameters on Functional capacity:Agility-motor coordination | up to 36 weeks
  Consist in a Standardized field test battery including:
  3.Agility-motor coordination (seconds)
Assessed changes from Baseline Physical Health Parameters on Functional capacity: Flexibility | up to 36 weeks
  Consist in a Standardized field test battery including:
  4.Flexibility (centimetres)
Assessed changes from Baseline Physical Health Parameters on Functional capacity: Handgrip strength | up to 36 weeks
  Consist in a Standardized field test battery including:
  5.Handgrip strength (kilograms)
Assessed changes from Baseline Incremental Exercise test: | up to 36 weeks
  All subjects performed a graded exercise test on a treadmill (Lode Valiant, Groningen, Netherlands) until exhaustion. Specifically, a modified Bruce protocol previously used in a similar sample and designed for a geriatric population. Participants were asked if they had ever walking on a treadmill and instructed of the incremental test. If necessary, we familiarized them with the treadmill by walking slowly until the initial protocol speed was achieved. Before start, subjects were instructed not to talk during the test because this is known to affect the breathing and gas exchange. Participants began walking to 2.7 km/h at 0% inclination grade, every 2 minutes the speed or/and inclination were increased according the modified Bruce protocol. VO2peak was considered as the highest observed value of oxygen consumption obtained in the last three intervals of 10 seconds.
Assessed changes from Baseline Physical Health by the Scale of instrumental activities of the daily life of Lawton and Brody | up to 36 weeks
  This scale measures the possibility of carrying out daily instrumental activities in daily life (Total score 0 to 8; higher value for better outcome).
Assessed changes from Baseline Physical Health of hemodynamic status | up to 36 weeks
  the hemodynamic status will be measured twice after 5 minutes at rest using a upper blood pressure monitor (M6 Omron):
  1. -Systolic and diastolic Blood pressure (mmHg)
  2. - Resting heart rate (beats per minute)
Assessed changes from Baseline Physical Health of Body Composition: Weight | up to 36 weeks
  Body Composition will be measured using a bio-impedanciometer (BIA; Tanita-MC-780MA MF 8-elc) including:
  1.Weight (in kilograms)
Assessed changes from Baseline Physical Health of Body Composition:Height | up to 36 weeks
  Body Composition will be measured using a Stadiometer (SECA):
  2.Height (in meters)
Assessed changes from Baseline Physical Health of Body Composition: Waist Circumference | up to 36 weeks
  Body Composition will be measured using an anthopometric flexible tape (SECA):
  3.Waist circumference (in centimetres)
Assessed changes from Baseline Physical Health of Body Composition: Body mass index | up to 36 weeks
  Body Composition will be measured as:
  4.Calculated body mass index (weight and height will be combined to report BMI in kg/m^2)
Assessed changes from Baseline Physical Health of Body Composition: Total body fluids | up to 36 weeks
  Body Composition will be measured using a bio-impedanciometer (BIA; Tanita-MC-780MA MF 8-elc) including:
  5. Total body fluids (litres).
Assessed changes from Baseline Blood Sample of the Cardio-metabolic Risk Factors Profile: Glucose. | up to 36 weeks
  The Cardio-metabolic Risk Factors Profile will be measured by several biochemical parameters including:
  1.Glucose (mg/dl)
Assessed changes from Baseline Blood Sample of the Cardio-metabolic Risk Factors Profile:Total cholesterol | up to 36 weeks
  The Cardio-metabolic Risk Factors Profile will be measured by several biochemical parameters including:
  2.Total cholesterol (mg/dl)
Assessed changes from Baseline Blood Sample of the Cardio-metabolic Risk Factors Profile:HDL cholesterol | up to 36 weeks
  The Cardio-metabolic Risk Factors Profile will be measured by several biochemical parameters including:
  3.HDL cholesterol (mg/dl)
Assessed changes from Baseline Blood Sample of the Cardio-metabolic Risk Factors Profile: LDL Cholesterol | up to 36 weeks
  The Cardio-metabolic Risk Factors Profile will be measured by several biochemical parameters including:
  4.LDL cholesterol (mg/dl)
Assessed changes from Baseline Blood Sample of the Cardio-metabolic Risk Factors Profile:triglycerides | up to 36 weeks
  The Cardio-metabolic Risk Factors Profile will be measured by several biochemical parameters including:
  5.triglycerides (mg/dl)
Assessed changes from Baseline Blood Sample of the Cardio-metabolic Risk Factors Profile:Apolipoprotein B | up to 36 weeks
  The Cardio-metabolic Risk Factors Profile will be measured by several biochemical parameters including:
  6.Apolipoprotein B (g/l)
Assessed changes from Baseline Blood Sample of the Cardio-metabolic Risk Factors Profile:Insulin | up to 36 weeks
  The Cardio-metabolic Risk Factors Profile will be measured by several biochemical parameters including:
  7.Insulin (μlU/mL)
Assessed changes from Baseline Blood Sample of the Cardio-metabolic Risk Factors Profile: HOMA | up to 36 weeks
  The Cardio-metabolic Risk Factors Profile will be measured by several biochemical parameters including:
  8.Insulin resistance (HOMA is calculated as fasting insulin [pmol/l]/6.945).
Assessed changes from Baseline Blood Sample of the Antioxidant Capacity | up to 36 weeks
  The Antioxidant Capacity will be measured by the following markers:
  1. - The 2,2'-azino-bis-3-ethylbenzthiazoline-6-sulphonic acid (ABTS)
  2. Oxygen radical absorption capacity (micromol/100 milliliter)
  3. Ferric reducing antioxidant potential (mmol/l).
Assessed changes from Baseline Blood Sample of the Neurotrophic Factor Derived from the Brain (neurotransmitter) | up to 36 weeks
  The Neurotrophic Factor Derived from the Brain will be measured as followed:
  1.-The brain-derived neurotrophic factor (BDNF in ug/L) will be measured in serum using the ELISA Kit (Enzyme-linkerd immunosorbent Assay) of RAyBio Human BDNF (RAFER). This marker is highly related to brain function and could mediate or explain to a certain extent the results of the EFICCOM project.
Assessed of Baseline levels for Cerebrospinal fluid: | baseline
  The Cerebrospinal fluid will be measured as followed:
  1.- Lumbar punctures will be performed accordinly with clinical standards and procedures manual at the specific unit of Neurology from the Puerta del Mar Hospital. CSF samples will be frozen on dry-ice soon after collection (~1 hour) and shipped to the university unit responsible for the analysis. This marker is highly relevant for the identifciation of the real risk for mild cognitive impairment using gold standard biomarkers of the EFICCOM project.
Assessed changes from Baseline Quality of life as assessed through the quality of life questionnaire related to health (Short-Form Health Survey 36 -SF36) | up to 36 weeks
  The Short-Form Health Survey 36 -SF36 includes 8 dimensions scored from 0 to 100 (higher value for better outcome).
Assessed changes from Baseline of Depression using the Geriatric Depression Scale (GDS) | up to 36 weeks
  The Depression will be measured using the Geriatric Depression Scale-GDS which is composed of 15 questions with dichotomous answers (yes / no) specifically designed for the elderly population and will be used to rule out depression. The GDS score from 0 to 15, where higher value means a worse outcome.
Assessed changes from Baseline of Sociodemographic Characteristics: Age. | up to 36 weeks
  The Sociodemographic Characteristics will be measured by several items including:
  1. Age (years)
Assessed changes from Baseline of Sociodemographic Characteristics.Sex. | up to 36 weeks
  The Sociodemographic Characteristics will be measured by several items including:
  2. Sex (male or female)
Assessed changes from Baseline of Sociodemographic Characteristics.Marital Status. | up to 36 weeks
  The Sociodemographic Characteristics will be measured by several items including:
  3.Marital status (Categorical variable: Single, Married or with a partner, Widowed and without partner, legally separated or divorced)
Assessed changes from Baseline of Sociodemographic Characteristics.Educational level and socio-economic status. | up to 36 weeks
  The Sociodemographic Characteristics will be measured by several items including:
  4. Educational level and socio-economic status (Ordinal variables where the higher the better: low, middle, high for Educational level; Low and high for socio-economic status)
Assessed changes from Baseline of Sociodemographic Characteristics.Family history of dementia. | up to 36 weeks
  The Sociodemographic Characteristics will be measured by several items including:
  5.Family history of dementia (yes/no and details),
Assessed changes from Baseline of Sociodemographic Characteristics.Medication. | up to 36 weeks
  The Sociodemographic Characteristics will be measured by several items including:
  6.Number and type of Medications (register)
Assessed changes from Baseline of Sociodemographic Characteristics. Other pathologies. | up to 36 weeks
  The Sociodemographic Characteristics will be measured by several items including:
  7.Presence of other pathologies (list of diseases).

CONTACTS AND LOCATIONS:
Overall Officials: David Jiménez Pavón, PhD, Principal Investigator — University of Cádiz
Locations (1):
- University of Cádiz, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Velazquez-Diaz D, Cadenas-Sanchez C, Molina-Guzman FA, Saenz-Carrasco JA, Gonzalez-Rosa JJ, Erickson KI, Carbonell-Baeza A, Jimenez-Pavon D. A new set of estimated cardiorespiratory fitness equations are associated with cognitive performance in older adults. Geroscience. 2023 Jun;45(3):1649-1666. doi: 10.1007/s11357-022-00718-w. Epub 2023 Jan 19. PMID 36653578
- See also: This is the website of the current project — http://eficcom.uca.es/